CLINICAL TRIAL: NCT03650803
Title: Role of Magnetic Resonance Fingerprinting and Quantitative MR Imaging in Assessment of Response to Neo-Adjuvant Chemotherapy in Breast Cancer
Brief Title: Role of Magnetic Resonance Fingerprinting and Quantitative MR Imaging in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CASE3118
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: 3D MR Fingerprinting; Quantitative MR Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 3D MR Fingerprinting scan (Experimental): Three separate 3D MR fingerprinting scans: Before the start of chemotherapy, 7-10 days after the first cycle of chemotherapy, and within 1 month of the end of chemotherapy treatment.
  Interventions: Device: 3D MR Fingerprinting scan

INTERVENTIONS:
Device: 3D MR Fingerprinting scan — 3D MR Fingerprinting technique is a non-contrast technique and generates quantitative information about MR-visible tumors without having to administer contrast.
  MR Fingerprinting software is used in conjunction with a standard-of-care MRI scan.

SUMMARY:
The purpose of this study is to determine if new methods of MRI imaging can better measure participants' response to chemotherapy treatment.

DETAILED DESCRIPTION:
The objectives of this study are to assess the utility of quantitative Magnetic Resonance Imaging (MRI) in assessment of response to neo-adjuvant chemotherapy in breast cancer. Magnetic Resonance (MR) Fingerprinting based relaxometry allows quantification of T1 and T2 relaxation times of tumor and normal breast tissue. Response to chemotherapy is associated with measurable changes in these properties and may be used to predict treatment response earlier than conventional MRI. The study team hypothesize that 3D MRF before, during and after chemotherapy can provide additional quantitative information about changes during treatment and may predict early response to chemotherapy.

During visit 1, 3D MR Fingerprinting images will be added to the clinical MRI scan before start of chemotherapy. The additional research images will take less than 20 minutes to acquire During visit 2, patients will be scheduled for a research only non-contrast 3D MR Fingerprinting scan 7-10 days after the first cycle of chemotherapy. Acquisition of images will take approximately 30 minutes.

During visit 3, if the treating physician orders a clinical MRI scan within 1 month of the end of chemotherapy treatment, the investigators will add a 3D MR Fingerprinting sequence to the clinical scan. The additional research images will take less than 20 minutes to acquire. If the patient is not scheduled for a clinical scan within 1 month of the end of chemotherapy treatment, the investigators will contact the patient to schedule a research only 3D MR Fingerprinting scan. The study team would like to administer IV gadolinium contrast for research purposes. Patients will be reconsented prior to the research only scan to determine whether or not they will receive IV contrast. If the patient declines administration of contrast for the post treatment scan, the study team will perform a non-contrast scan. Acquisition of images will take 30-45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven cases of breast cancer

Exclusion Criteria:

* Patients with onlybenign lesion
* Patients with onlyductal carcinomain situ (DCIS)
* Patients with recurrent/ residual breast cancer in same breast
* Pregnant women
* Lactating Women6.Patients with ferromagnetic or otherwise non-MRI compatible aneurysm clips.
* The presence of an implanted medical device that is not MRI-compatible, including, but not limited to: pacemaker, defibrillator
* Patients with contraindications for MRIdue to embedded foreign metallic objects. Bullets, shrapnel, metalwork fragments, or other metallic material adds unnecessary risk to the patient.
* Known history of severe claustrophobia
* Patients under the age of 18
* For patients with known history of allergic reaction to MR contrast material or abnormal kidney function (GFR < 40 mL/ min), a contrast enhanced exam will not be performed; however, a non-contrast exam may be performed in these patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Marshall, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 3D MR Fingerprinting Scan: Three separate 3D MR fingerprinting scans: Before the start of chemotherapy, 7-10 days after the first cycle of chemotherapy, and within 1 month of the end of chemotherapy treatment.
  3D MR Fingerprinting scan: 3D MR Fingerprinting technique is a non-contrast technique and generates quantitative information about MR-visible tumors without having to administer contrast.
  MR Fingerprinting software is used in conjunction with a standard-of-care MRI scan.
Period: Overall Study
Arm/Group | 3D MR Fingerprinting Scan
Started | 14
Completed | 8
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | 3D MR Fingerprinting Scan
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 14
Pathology [Count of Participants; unit: Participants] — Invasive ductal carcinoma (IDC) was measured by the Nottingham Histologic Scoring System that takes three factors into consideration to tell whether a tumor is well, moderately or poorly differentiated. The three factors include gland formation (scored 1-3), nuclear pleomorphism (scored 1-3), and mitotic count (scored 1-3). A higher tumor grade usually indicates a poorer prognosis. Grading is as follows: Grade I: tumors with a total score of 3-5; Grade II: tumors with a total score of 6-7; Grade III: tumors with a total score of 8-9. Population: Population excludes 6 participants who were lost to follow-up.
  Participants
    number analyzed (Participants) | 8
    IDC Grade 2 | 2
    IDC Grade 3 | 6
Breast Parenchyma Composition [Count of Participants; unit: Participants] — Population: Population excludes 6 participants who were lost to follow-up.
  Participants
    number analyzed (Participants) | 8
    Fatty | 1
    Heterogeneously Dense | 3
    Dense | 0
    Extremely Dense | 4
Hormone Status [Count of Participants; unit: Participants] — Population: Population excludes 6 participants who were lost to follow-up.
  Participants
    number analyzed (Participants) | 8
    PPN | 2
    PNN | 1
    NNP | 2
    TN | 2
    PPP | 1

OUTCOME MEASURES:

1. Primary Outcome: Utility of Percentage Change in Longitudinal (T1) and Transverse (T2) Relaxation Times From Baseline to First Cycle of Treatment in Assessment of Response to Neo-adjuvant Chemotherapy in Breast Cancer.
Description: For each patient the first MRF scan was performed at the baseline before chemotherapy and the second MRF scan was performed 7-10 days after the first cycle of chemotherapy. Quantitative T1 and T2 relaxation times measured using MRF were used to characterize the breast lesions and predict the treatment response at an early phase (7-10 days after one-cycle of neoadjuvant chemotherapy).
  Changes in relaxation times (T1 or T2) between the baseline and 7-10 days after the first cycle of chemotherapy were used for predicting the early prediction of treatment response. Both T1 and T2 relaxation times were measured in the unit of millisecond. The unit of the measurement for this primary outcome was percentage changes of relaxation times (T1 or T2) obtained at the two different time points.
  The pathological results obtained after the breast surgery were used as the ground truth to determine patients response to the treatment and correlated with the findings obtained using MRF.
Time Frame: 2 years from start of study
Population: Only the participants who have completed at least the first two MRF scans were included in this data analysis. Six participants are excluded due to being lost to follow-up.
Measure: Mean (Standard Deviation); unit: Percentage change of relaxation time
Groups:
- Responders to 3D MR Fingerprinting Scan: Patients with biopsy proven cases of breast cancer who were scheduled to undergo chemotherapy treatment were enrolled in this study. Quantitative MRF scans were acquired at the baseline before the treatment, 7-10 days after the first cycle of chemotherapy, and at the end of treatment. All MRF scans were acquired without any contrast administration. Final surgico-pathology results would be used for response assessment. Pathology reports with pT0N0 would be designated as pathological complete response or Responder in this study.
- Non-Responders to 3D MR Fingerprinting Scan: Patients with biopsy proven cases of breast cancer who were scheduled to undergo chemotherapy treatment were enrolled in this study. Quantitative MRF scans were acquired at the baseline before the treatment, 7-10 days after the first cycle of chemotherapy, and at the end of treatment. All MRF scans were acquired without any contrast administration. Final surgico-pathology results would be used for response assessment. Presence of any residual tumor on pathology would be considered as Non-Responder in this study.
Arm/Group | Responders to 3D MR Fingerprinting Scan | Non-Responders to 3D MR Fingerprinting Scan
Number analyzed (Participants) | 3 | 5
Percentage change of relaxation time
  MRF T1 Changes | -19.8 (19.3) | 5.4 (9.9)
  MRF T2 Changes | -21.4 (4.2) | -7.1 (10.2)
Statistical Analysis 1: Comparison: Responders to 3D MR Fingerprinting Scan vs Non-Responders to 3D MR Fingerprinting Scan; MRF T1 Changes; Test type: Other — Significance (alpha) set to 0.05; p = 0.046, t-test, 1 sided
Statistical Analysis 2: Comparison: Responders to 3D MR Fingerprinting Scan vs Non-Responders to 3D MR Fingerprinting Scan; MRF T2 Changes; Test type: Other — Significance (alpha) set to 0.05; p = 0.064, t-test, 2 sided

2. Primary Outcome: Longitudinal Relaxation (T1) and Transverse Relaxation (T2) Times of Breast Tumor
Description: From the 3D MR Fingerprinting maps, T1 and T2 relaxation times will be obtained from breast tumors at the baseline condition before the treatment.
Time Frame: 2 years from start of study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Responders to 3D MR Fingerprinting Scan | Non-Responders to 3D MR Fingerprinting Scan
Number analyzed (Participants) | 3 | 5
milliseconds
  MRF T1 values before treatment | 1304.3 (121.5) | 1264.6 (266.6)
  MRF T2 values before treatment | 77.0 (6.6) | 68.8 (24.8)
Statistical Analysis 1: Comparison: Responders to 3D MR Fingerprinting Scan vs Non-Responders to 3D MR Fingerprinting Scan; MRF T1 relaxation time; Test type: Other — Significance (alpha) set to 0.05; p = 0.820, t-test, 2 sided
Statistical Analysis 2: Comparison: Responders to 3D MR Fingerprinting Scan vs Non-Responders to 3D MR Fingerprinting Scan; MRF T2 relaxation time; Test type: Other — Significance (alpha) set to 0.05; p = 0.605, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through study completion, up to 6 months for each enrolled patient.
Arm/Group | 3D MR Fingerprinting Scan
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3D MR Fingerprinting Scan (N=14)
Nervous system disorders, Other: MRI exacerbated pre-existing Menier's Disease (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/03/NCT03650803/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT03650803/ICF_001.pdf